CLINICAL TRIAL: NCT04656587
Title: Bilevel Positive Airway Pressure (BPAP) in Pediatric Asthma Exacerbations: A Pilot Study
Brief Title: BPAP in Pediatric Asthma Pilot Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution.
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAS8758
Record Dates: First submitted 2020-11-23; First posted 2020-12-07 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Asthma in Children; Status Asthmaticus
Keywords: non-invasive ventilation; BPAP; continous albuterol; pediatrics
MeSH Terms: conditions — Status Asthmaticus | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard Therapy (Control) (Other): Standard status asthmaticus therapy with continuous beta-agonist, steroids and oxygen as needed.
  Interventions: Other: Standard Therapy
- Standard Therapy plus BPAP (Experimental): Application of BPAP along with standard status asthmaticus therapy with continuous beta-agonist, steroids and oxygen as needed.
  Interventions: Device: Philips Respironics V60 Non-invasive ventilator, BPAP; Other: Standard Therapy

INTERVENTIONS:
Device: Philips Respironics V60 Non-invasive ventilator, BPAP — Continuous albuterol will be administered through the BPAP circuit.
  Other Names: Philips Respironics V60 Non-invasive ventilator
  Arms: Standard Therapy plus BPAP
Other: Standard Therapy — Standard status asthmaticus therapy with continuous beta-agonist, steroids and oxygen as needed.

SUMMARY:
The investigators aim to study the effect and safety of bilevel positive airway pressure (BPAP) in children with moderate to severe asthma exacerbations - by examining the effects of early initiation of BPAP in pediatric patients who present to the emergency room with a moderate to severe asthma exacerbation. The study is interested in how early initiation of BPAP affects PRAM scores, vital signs, as well as the total duration of continuous albuterol in the patient population.

DETAILED DESCRIPTION:
Asthma is the most common chronic illness of childhood. Bilevel positive airway pressure (BPAP) has been suggested as an adjunct therapy in the setting of moderate to severe asthma exacerbations. It is a form of noninvasive positive pressure ventilation that provides both an inspiratory positive airway pressure (IPAP) as well as an expiratory positive airway pressure (EPAP).

The goal of this study is to determine the feasibility of enrolling, randomizing, and completing data collection in at least 30 participants over a one-year period. The investigators will enroll children 5 to 17 years of age presenting to the emergency department with a moderate to severe asthma exacerbation. Eligible participants will be randomized into two groups: standard therapy (continuous albuterol) or standard therapy plus BPAP. The following data will be collected: Pediatric Respiratory Assessment Measure (PRAM) score at 0, 2 and 4 hours, vital signs at 0, 2 and 4 hours, rate of adverse events and Pediatric Intensive Care Unit (PICU) admissions, duration continuous albuterol, length of hospital stay, and rates of intubations or deaths.

ELIGIBILITY:
Inclusion Criteria:

* 5 to 17 years of age (inclusive) presenting to the Emergency Department (ED) with an asthma exacerbation
* Prior clinician diagnosis of asthma
* PRAM score of 4 or greater after initial albuterol/atrovent back to backs, steroids, +/- oxygen
* Need for continuous nebulized albuterol therapy

Exclusion Criteria:

* Hypercapneic respiratory failure (partial pressure of carbon dioxide > 60 mmHg)
* Hypoxemic respiratory failure (SaO2 < 90% with fraction of inspired oxygen > 0.35)
* Presence of a tracheostomy or baseline noninvasive ventilation requirement
* Non-asthma causes of wheezing (foreign body, tracheomalacia, vocal cord dysfunction, pulmonary edema, uncorrected congenital heart disease, cystic fibrosis)
* Contra-indication to BPAP (facial trauma, uncontrollable vomiting, hypotension for age, Glasgow Coma Scale (GCS) 8 or less, drowsiness or confusion, known or clinical suspicion for pneumothorax, pneumomediastinum, or subcutaneous emphysema, pregnancy, current weight < 20kg)

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Feasibility of successfully enrolling, randomizing, and completing data collection in 30 participants within one year. | One year
  Feasibility defined as successfully enrolling, randomizing, and completing data collection in 30 participants within one year in the pediatric emergency department.

SECONDARY OUTCOMES:
Difference in PRAM Score | At 2 and 4 hour time points
  Difference in PRAM scores at 2 and 4 hours. PRAM scores range from 0 to 12 with a score of 4 or greater indicating moderate to severe disease. Decreasing scores reflect clinical improvement in response to therapy.
Difference in Respiratory Rate | At 2 and 4 hour time points
  Difference in respiratory rate measured in breaths per minute (bpm).
Difference in Oxygen Saturation | At 2 and 4 hour time points
  Difference in percent oxygen saturation.
Difference in Heart Rate | At 2 and 4 hour time points
  Difference in heart rate measured in beats per minute (bpm).
Difference in Systolic and Diastolic Blood Pressure | At 2 and 4 hour time points
  Difference in systolic and diastolic blood pressure measured in millimeters of mercury (mmHg).
Difference in Duration of continuous beta-agonist therapy | Until therapy is completed, approximately 24 hours
  Difference in duration of continuous beta-agonist therapy measured in hours.
Rate of PICU Admission | Until hospital discharge, approximately 2 days
  Rate of admissions from the Emergency Department (ED) to PICU versus home or to the pediatric floor
Length of Stay | Until hospital discharge, approximately 2 days
  Length of stay, measured in days, in the ED, PICU, or hospital

OTHER OUTCOMES:
Cumulative Number of Adverse Events | Until hospital discharge, approximately 2 days
  The total number of adverse events per arm will be reported. Adverse events include air leak syndrome, aspiration pneumonia, skin break down, hypotension, intubation, death or other adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick T Wilson, MD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Korang SK, Baker M, Feinberg J, Newth CJ, Khemani RG, Jakobsen JC. Non-invasive positive pressure ventilation for acute asthma in children. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD012067. doi: 10.1002/14651858.CD012067.pub3. PMID 39356050